CLINICAL TRIAL: NCT00263263
Title: Phase 2 Randomized Double-Blind Comparison of Sirolimus-Eluting Stent Versus Bare-Metal Stent Implantation in Degenerated Saphenous Vein Grafts
Brief Title: RRISC Study: Reduction of Restenosis In Saphenous Vein Grafts With Cypher Sirolimus-Eluting Stent.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antwerp Cardiovascular Institute Middelheim (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCUBATE-001
Record Dates: First submitted 2005-12-07; First posted 2005-12-08 (Estimated); Last update posted 2007-03-14 (Estimated); Status verified 2007-03

CONDITIONS: Stable Angina; Unstable Angina; Coronary Artery Disease; Saphenous Vein Graft Disease
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: sirolimus-eluting stent
Device: bare metal stent

SUMMARY:
Context: Sirolimus-eluting-stents have improved the benefits of percutaneous interventions in native coronary arteries reducing the occurrence of restenosis and repeated revascularization, however saphenous vein grafts have been always excluded form randomized trials.

Objective: To evaluate the angiographic and clinical impact of sirolimus-eluting-stents with respect to bare-metal-stents in degenerated vein grafts.

Design: Double-blind randomized controlled non-industry-sponsored trial.

Setting: A single-center tertiary-care referral hospital.

Patients: All patients are randomly allocated to sirolimus-eluting-stent implantation or the corresponding bare-metal-stent. All patients are followed clinically and repeated angiographic follow-up is performed in all at 6-months.

Main outcome measure: Primary end-point is 6-months angiographic in-stent late loss. Secondary end-points include: binary angiographic in-stent and in-segment restenosis, intravascular-ultrasound-measured neo-intimal hyperplasia volume and all the clinical events (death, myocardial infarction, target-lesion and target-vessel revascularization).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years-old
* clear signs and/or symptoms of stable or unstable angina or documented silent ischemia
* one or more de-novo target lesions (>50% diameter stenosis by visual estimate) localized in one or more diseased SVG with a reference vessel diameter (RVD) included between 2.5 and 4.0 mm (by visual estimate)
* signed informed consent.

Exclusion Criteria:

* Myocardial Infarction within the previous 7 days
* documented left ventricular ejection fraction <25%
* impaired renal function (creatinine >3.0 mg/dl) at the time of treatment
* outflow obstruction of the graft due to distal anastomotic stenosis
* totally occluded Saphenous Vein Graft
* brachytherapy treatment in the index vessel before enrollment
* life expectancy less than 12 months
* known allergy to aspirin, clopidogrel bisulfate, heparin, stainless steel, contrast agent or sirolimus
* hemorrhagic diatheses
* a recent positive pregnancy test, breast-feeding, or the possibility of a future pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2003-09; Study Completion 2005-12

PRIMARY OUTCOMES:
In-stent late loss

SECONDARY OUTCOMES:
in-segment late loss
binary angiographic in-stent restenosis
binary angiographic in-segment restenosis
intravascular-ultrasound-measured neo-intimal hyperplasia volume
death
myocardial infarction
target-lesion revascularization
target-vessel revascularization
stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Vermeersch, MD, Principal Investigator — Antwerp Cardiovascular Institute Middelheim; Glenn Vanlangenhove, MD, PhD, Study Chair — Antwerp Cardiovascular Institute Middelheim; Pierfrancesco Agostoni, MD, Study Director — Antwerp Cardiovascular Institute Middelheim
Locations (1):
- Antwerp Cardiovascular Institute Middelheim, Antwerp, Belgium

REFERENCES:
- [Derived] Vermeersch P, Agostoni P, Verheye S, Van den Heuvel P, Convens C, Van den Branden F, Van Langenhove G; DELAYED RRISC (Death and Events at Long-term follow-up AnalYsis: Extended Duration of the Reduction of Restenosis In Saphenous vein grafts with Cypher stent) Investigators. Increased late mortality after sirolimus-eluting stents versus bare-metal stents in diseased saphenous vein grafts: results from the randomized DELAYED RRISC Trial. J Am Coll Cardiol. 2007 Jul 17;50(3):261-7. doi: 10.1016/j.jacc.2007.05.010. Epub 2007 Jun 13. PMID 17631219
- [Derived] Vermeersch P, Agostoni P, Verheye S, Van den Heuvel P, Convens C, Bruining N, Van den Branden F, Van Langenhove G. Randomized double-blind comparison of sirolimus-eluting stent versus bare-metal stent implantation in diseased saphenous vein grafts: six-month angiographic, intravascular ultrasound, and clinical follow-up of the RRISC Trial. J Am Coll Cardiol. 2006 Dec 19;48(12):2423-31. doi: 10.1016/j.jacc.2006.09.021. Epub 2006 Nov 28. PMID 17174178